CLINICAL TRIAL: NCT05002400
Title: Evaluation of the PS100B for the Diagnostic of Stroke With Patients Out of Delay for Thrombolysis or Thrombectomy
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STROkE
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: PS100B; stroke; out of delay; diagnostic
MeSH Terms: conditions — Stroke; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample in order to measure the value of PS100B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Numerous patients are addressed to the Emergency Department for unspecific symptoms which can evoke a stroke, such as vertigo, isolated motor deficit, behavior disorder.

For these patients, when they arrive out of time for specific treatments such as thrombolysis and thrombectomy, the cerebral imagery is not an emergency, but necessary to confirm or invalidate the diagnostic of stroke.

If a biomarker could exclude the diagnostic of stroke, we could avoid an imagery for these patients.

PS100B is a biomarker whose blood level increases in case of stroke. It has already proven a prognostic value. Until now, it hasn't proven a diagnostic value because it take a few hours to increase in the blood.

It could have in prognostic value for patients who have the symptoms for more than 24 hours.

STROkE is a diagnostic, prospective, monocentric study, conducted at University Hospital Center of Poitiers (France).

The aim is to determine the value of PS100B to exclude the diagnostic of a stroke in case of evocative symptoms, for patients who are out of delay for a thrombolysis or a thrombectomy.

Patients eligible are the ones who present to the emergency department with symptoms evocative of stroke for more than 24 hours and less than 4 days. Patients included have a sample of blood withdrawn, in order to measure PS100B blood level.

The diagnostic of stroke is than confirmed or excluded by an adjudication comity, who are unaware of the result of PS100B blood level.

The diagnostic value of PS100B is determined with the help of a ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the Emergency Department of the University Hospital Center of Poitiers for the following symptoms, which last since more then 24 hours et less then 4 days :
* sensitive or motor deficit of one or several limbs
* facial paralysis
* impairment of speech
* dysarthria
* vertigo
* impairment of vision
* oculomotor disorder
* diplopia
* free patient, without guardianship or curatorship, or subordination
* patient not objecting to research

Exclusion Criteria:

* head trauma that occured less then 15 days ago
* known cerebral mass or melanoma
* refusal to participate in research
* patient benefiting from enhanced protection, namely: minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection
* pregnant and/or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the Emergency Department of the University Hospital Center of Poitiers for symptoms evocative of stroke for more then 24 hours and less then 4 days, that fit the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of PS100B | 1 day
  Determine the best couple sensibility / specificity of the blood value of PS100B with the help of a Receive Operating Charasteristics (ROC) curve for patients who present with symptoms evocative of stroke since more than 24 hours and less than 4 days

SECONDARY OUTCOMES:
Value of PS100B for ischemic strokes and hemorrhagic strokes | 1 day
  Comparison of the mean value of PS100B between patients with ischemic strokes and hemorrhagic strokes
Value of PS100B and time delay since the beginning of the symptoms | 1 day
  Stratification of the value of PS100B with the delay of apparition of the symptoms and realization of the blood sample
Prognostic value of PS100B | 28 days
  Comparison of the value of PS100B and the patient's outcomes 28 days after inclusion. The patient's outcome will be assessed as follow : hospitalization, death and self-rated health perception.
  The self-rated health perception will be assessed with the scale EuroQOL (EQ)-5D-5L. The scale EQ-5D-5L is composed of :
  * a score on 5 levels : from 1 to 3 (no problem) and 4 to 5 (with problems)
  * analogic scale from 0 to 100 (0 = worst health perception ; 100 = best health perception)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Henri MONDOR, Créteil
  - C.H.U. de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided